CLINICAL TRIAL: NCT05043363
Title: LumenEye During CovID-19 (LuCID Study)
Brief Title: LuCID - Investigating the Use of a Novel Digital Rectoscope for Community Examinations During COVID-19
Acronym: LuCID
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 285758
Record Dates: First submitted 2021-09-13; First posted 2021-09-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Bowel Cancer; Bowel Diseases, Inflammatory; Rectal Bleeding
Keywords: endoscopy; digital; examination; primary care
MeSH Terms: conditions — Intestinal Neoplasms; Inflammatory Bowel Diseases; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: 1. Patients with an established diagnosis of inflammatory bowel disease who have been identified as being 'at risk' by either their secondary care doctor or GP and now require endoscopic assessment for ongoing disease symptoms but are unable to access endoscopy services urgently.
  2. Patients presenting directly to their GP practice with symptoms of anorectal disease (e.g. rectal bleeding or pain) or symptoms that would warrant referral to a hospital under a 2WW appointment according to NICE criteria
  Recruited patients will undergo rectal examination in primary care with the LumenEye X1 with either contemporaneous or retrospective image review by a secondary care clinician. This will require a glycerine suppository to be administered. Patient feedback will be sought with a post-procedural questionnaire.
  Interventions: Device: LumenEye X1 digital rectoscope

INTERVENTIONS:
Device: LumenEye X1 digital rectoscope — The LumenEye X1 is a novel digital rectoscope that introduces digital HD imaging and improved ergonomics to conventional rigid sigmoidoscopy.

SUMMARY:
The LumenEye scope and CHiP platform will be piloted in a number of clinical settings including remote colorectal clinics. The rationale is to perform an initial pilot study to determine the clinical utility of the LumenEye device for use in primary and secondary care settings.

The main hypothesis is that digital rectoscopy is safe and acceptable to clinicians including general practitioners and can significantly reduce the burden of endoscopy referral to and within secondary care centres.

DETAILED DESCRIPTION:
All clinicians performing investigations with the LumenEye will undergo training and quality assurance assessment. The first 5 procedures will be performed with a proctor to ensure that this is performed safely using appropriate PPE according to Public Health England Recommendations.

The primary study site will be based at Imperial College NHS trust which is a recognized National Bowel Cancer Screening (NBCS) Centre of excellence. The Imperial endoscopy suite performs over 10,000 endoscopic procedures each year.

All patients enrolled into the study will be asked to have a glycerine suppository prior to the examination. They will be examined by the primary care physician in the clinic as per a standard rigid sigmoidoscopy assessment. Physicians may take biopsies if required but only if the physician feels this is warranted for clinical use. There is no requirement for research specimens in this study.

All doctors using the LumenEye will asked to record images showing standard anatomical locations including:

1. The rectosigmoid junction
2. Each rectal haustral fold
3. Exit from the rectum. Videos will also be recorded for any pathology identified. Virtual clinics will be coordinated by the CI and Co-Is. During these clinics, a secondary care physician or surgeon will be available to discuss the case with the GP. These could be performed in real time with the patient present during a live examination or they could be performed retrospectively as part of a multidisciplinary team meeting.

Clinicians will be asked to provide qualitative feedback data with each use concerning device performance. This will be in the form of a short questionnaire, split into technical performance, views achieved, diagnostic yield, quality of the telemedicine interaction, patient outcome (discharged or referred to formal endoscopy) and adverse events.

Patient feedback will be requested through a validated questionnaire.. All clinicians providing advice and guidance via CHiP will be asked to provide data on the quality of the views, the stability of the platform and to provide information on the diagnosis. All data pertaining to follow up colonoscopy or flexible sigmoidoscopy will be used as a comparator group for a diagnostic sensitivity / specificity analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Patients with any of the following:

  * Positive Faecal occult blood test / Faecal immunochemical test (FIT)
  * Positive faecal calprotectin.
  * Established history of polyps and/or adenomas
* 2WW patients referred to a colorectal clinic
* Known IBD patients with flare symptoms
* Patients with a suspected new diagnosis of IBD

Exclusion Criteria:

* Inability to consent
* Inability to communicate effectively in English
* Pregnancy
* Unfit for bowel preparation
* Anal stricture
* Allergy to plastic
* Inability to lie flat for more than 10 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified for recruitment via two routes:
  1. Patients with an established diagnosis of inflammatory bowel disease who have been identified as being 'at risk' by either their secondary care doctor or GP and now require endoscopic assessment for ongoing disease symptoms but are unable to access endoscopy services urgently.
  2. Patients presenting directly to their GP practice with symptoms of anorectal disease (e.g. rectal bleeding or pain) or symptoms that would warrant referral to a hospital under a 2WW appointment according to NICE criteria
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is undecided

REFERENCES:
- [Result] Lewis J, Askari A, Mehta A, Razak Y, Patel P, Misra R, Tilney H, Ahmed T, Ahmed M, Syeed A, Camilleri-Brennan J, Nicholls RJ, Kinross JM. A novel digital rectoscope for the triage of lower gastrointestinal symptoms in primary care: a prospective multicentre feasibility study. BJGP Open. 2022 Sep 28;6(3):BJGPO.2022.0036. doi: 10.3399/BJGPO.2022.0036. Print 2022 Sep. PMID 35728817

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from general practice or from urgent suspected colorectal cancer referral waiting lists held in secondary care. 114 patients were enrolled in the study from five NHS regions between November 2020 and June 2021.
Pre-assignment Details: This was an observational feasibility study with no exclusions after recruitment.
Groups:
- Observational Cohort: 1. Patients with an established diagnosis of inflammatory bowel disease who have been identified as being 'at risk' by either their secondary care doctor or GP and now require endoscopic assessment for ongoing disease symptoms but are unable to access endoscopy services urgently.
  2. Patients presenting directly to their GP practice with symptoms of anorectal disease (e.g. rectal bleeding or pain) or symptoms that would warrant referral to a hospital under a 2WW appointment according to NICE criteria
  Recruited patients will undergo rectal examination in primary care with the LumenEye X1 with either contemporaneous or retrospective image review by a secondary care clinician. This will require a glycerine suppository to be administered. Patient feedback will be sought with a post-procedural questionnaire.
  LumenEye X1 digital rectoscope: The LumenEye X1 is a novel digital rectoscope that introduces digital HD imaging and improved ergonomics to conventional rigid sigmoidoscopy.
Period: Overall Study
Arm/Group | Observational Cohort
Started | 114 (November 2020)
Completed | 110 (June 2021)
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Observational Cohort: 1. Patients with an established diagnosis of inflammatory bowel disease who have been identified as being 'at risk' by either their secondary care doctor or GP and now require endoscopic assessment for ongoing disease symptoms but are unable to access endoscopy services urgently.
  2. Patients presenting directly to their GP practice with symptoms of anorectal disease (e.g. rectal bleeding or pain) or symptoms that would warrant referral to a hospital under a 2WW appointment according to NICE criteria
Arm/Group | Observational Cohort
Number analyzed (Participants) | 114
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [36 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Experience of LumenEye Examination
Description: Assessing the percentage of participants with positive responses to the patient experience questionnaire, which is answered with a 5 point Likert scale
Time Frame: On the day of examination
Measure: Number; unit: percentage of participants
Arm/Group | Observational Cohort
Number analyzed (Participants) | 110
percentage of participants
  Examination was more comfortable than expected | 75
  Examination more comfortable than previous rigid sigmoidoscopy | 67
  Examination in the community more convenient than in hospital | 95
  Sharing over images over CHiP is beneficial to care | 94
  Comfortable with sharing of images with secondary care | 97
  Reassured that images are reviewed by secondary care | 98

2. Primary Outcome: Clinician Experience of LumenEye Examination
Description: Assessing the the positive response rate by examining clinicians to their overall experience and certainty of diagnosis for each examination
Time Frame: On the day of examination
Population: Clinician reports on each examination
Measure: Number; unit: percentage of clinician experience
Arm/Group | Observational Cohort
Number analyzed (Participants) | 110
percentage of clinician experience
  Very confident in suspected diagnosis | 56
  Reasonably confident in suspected diagnosis | 35
  Visualisation of rectosigmoid junction with LumenEye | 89

3. Secondary Outcome: Diagnostic Accuracy of the LumenEye for the Detection of Rectal Pathology Including Tumour, Polyps and Inflammation
Description: To provide pilot data within the small study for the diagnostic accuracy of the LumenEye system as compared to conventional flexible endoscopy.
Time Frame: Diagnostic accuracy of the LumenEye examination to be compared with subsequent investigations completed by the time of analysis (2-9 months after study examination).
Population: Patients undergoing colonoscopy, flexible sigmoidoscopy, or CTVC after LumenEye examination.
Measure: Number; unit: Percent
Arm/Group | Observational Cohort
Number analyzed (Participants) | 48
Percent
  Sensitivity for diagnosis of tumour, polyp or inflammation | 90.0
  Specificity for diagnosis of tumour, polyp or inflammation | 88.9

ADVERSE EVENTS:
Time Frame: Adverse events were recorded and reported if occurring at the time of examination. Any delayed reports of adverse events were reported and recorded at the time of follow up to review the results of any subsequent investigations (this ranges from 9 months for the earliest participants to 2 months for the last participants).
Description: Any adverse events were to be reported at the time of examination.
Arm/Group | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT05043363/Prot_SAP_000.pdf